CLINICAL TRIAL: NCT00661310
Title: Optimizing Drug-Therapy in Patients, 80 Years and Older, in Order to Reduce Drug-Related Morbidity and Usage of Secondary Care - a Randomized Controlled Trial
Brief Title: Optimizing Drug-Therapy in Patients 80 Years and Older
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Henrik Toss, MD, PhD, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Uppsala80
Record Dates: First submitted 2008-04-14; First posted 2008-04-18 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-10

CONDITIONS: Drug-Related Problems
Keywords: re-admissions; medicines; management; patients; 80 years and older; acute; admissions; hospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Intervention by team consisting of Doctor, pharmacist and nurse
  Interventions: Other: Drug review 80+ -To reduce usage of hospital care
- C (No Intervention)

INTERVENTIONS:
Other: Drug review 80+ -To reduce usage of hospital care — drug review performed by multiprofessional team, including clinical pharmacist, in order to optimize drug therapy and reduce usage of hospital care. Also patient education and follow-up
  Arms: I

SUMMARY:
The purpose of this study is to measure the effects of an enhanced service where a pharmacists is part of the healthcare team on the ward (focusing on drug-related problems and transferring information between primary and secondary care). Primary outcome measure is visits to hospital during a 12-month follow-up period, and the population is patients 80 years and older.

DETAILED DESCRIPTION:
Optimising drug-therapy for patients, 80 years and older, to reduce hospital visits

Background and Objective:

Results from a pilot-study performed in 2004 at the Academic Hospital, Uppsala, including 214 consecutive patients (80 years old or older) showed that 9.4%-13.6% of the patients were acutely admitted to hospital due to a drug related problem1. Other similar international studies show that the frequency of drug-related hospital admissions stands for at least 14% of the acute admissions (14%-30.4%). Of these admissions it was estimated that 32%-69% were preventable 2,3,4.

A study from Antrim Hospital, Northern Ireland, showed that pharmacists´ involvement in the health care team can reduce the number of acute hospital admissions and improve quality of drug use5.

In view of these findings this study was initiated in 2005 with fundings from the Drug and Therapeutics committee, the County Council of Uppsala, the Division of Acute-Medicine and the Pharmacy Department at the Academic Hospital in Uppsala

Aim and objectives:

The Study Aim was to optimize drug-prescribing and drug use for patients 80 years and older.

The main objective was to reduce the number of hospital visits for patients 80-years old or older.

Design:

A randomized, controlled trial including 400 patients (200+200). Patients in the intervention group (I) received a patient interview on admission, drug counseling on discharge and a drug review - all performed by a clinical pharmacist. Patients in the control group (C) received standard care, without pharmacists´ involvement.

Patients were included between Oct 2005 and June 2006.

Setting:

Two wards at the Division of Acute-Medicine at Uppsala University Hospital, Sweden

Main Outcome Measures:

1) Frequency of hospital visits 12 months after (last included patient) discharge from hospital for (I) and (C).

ELIGIBILITY:
Inclusion Criteria:

* 80 years and older
* Acute admission to study ward

Exclusion Criteria:

* <80 years
* Scheduled admission
* Previously admitted to studyward during study period

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2005-09; Primary Completion 2006-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Effects on hospital visits | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Toss, MD PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Gillespie U, Alassaad A, Henrohn D, Garmo H, Hammarlund-Udenaes M, Toss H, Kettis-Lindblad A, Melhus H, Morlin C. A comprehensive pharmacist intervention to reduce morbidity in patients 80 years or older: a randomized controlled trial. Arch Intern Med. 2009 May 11;169(9):894-900. doi: 10.1001/archinternmed.2009.71. PMID 19433702